CLINICAL TRIAL: NCT07164053
Title: Image Quality Evaluation of Surgical Visualization Headset (Leica MyVeo) During Standard of Care Procedure Per User Manual
Brief Title: Evaluation of Image Quality and Safety of the MyVeo Surgical Visualization Headset During Standard Neurosurgical and Reconstructive Procedures Using Compatible Microscopes.
Acronym: IMED-MYVEO
Status: Not yet recruiting | Type: Observational
Sponsor: Leica Microsystems (Schweiz) AG (Industry)
Responsible Party: Sponsor
Other Study IDs: MYVEO-PMCFSTUDYPLAN-202501
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: High-Grade Glioma (WHO III-IV); Cerebral Vascular Conditions Requiring Surgical Intervention; Conditions Requiring Plastic and Reconstructive Surgery
Keywords: Surgical Visualization Headset; MyVeo; ARveo8x Microscope; Image Quality Assessment; Fluorescence Imaging; White Light Imaging; Neurosurgery; High-Grade Glioma; WHO Grade III-IV Glioma; Indocyanine Green (ICG); 5-Aminolevulinic Acid (5-ALA); GLOW400; GLOW800; Post-Market Clinical Follow-Up (PMCF); Head-Mounted Display (HMD); Stereoscopic 3D Imaging; Surgical Ergonomics; Surgical Workflow; Intraoperative Visualization; Digital Surgical Accessory
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MyVeo is an all-in-one surgical visualization headset used with compatible surgical microscopes and other medical imaging systems in the area of neurosurgery, ENT, spine, plastic and reconstructive su — MyVeo is an all-in-one surgical visualization headset used with compatible surgical microscopes (ARveo 8/ARveo 8x) and other medical imaging systems. It is a digital accessory to an operating surgical microscope that enables the visualization of the surgical field through a visualization headset including:
  * Display of surgical field illuminated and magnified by the surgical microscope (White Light).
  * Display of fluorescence of fluorophores within the indicated excitation and emission ranges, as defined by the respective filters (accessories to the compatible surgical microscopes ARveo 8x such as GLOW400 and GLOW800).

SUMMARY:
This study looks at how well the MyVeo surgical visualization headset works during routine surgeries. MyVeo is a wearable device that helps surgeons see the surgical area in high detail, including blood flow and tissue fluorescence, without needing to look through a traditional microscope. The study will involve patients undergoing brain, spine, ENT, or reconstructive surgery, where MyVeo is used as part of the standard care. Surgeons will rate the image quality, comfort, and safety of using MyVeo. The goal is to confirm that MyVeo provides clear images and supports safe and effective surgery. No extra procedures or risks are added for patients.

ELIGIBILITY:
Inclusion Criteria:

Candidates for the IMED-MyVeo study protocol must be appropriate patients for the applicable indication of use and have to fulfil the following inclusion criteria to be eligible for the recruitment of the study.

1. Participants must be 18 years of age or older at the time of signing the informed consent.
2. The participant or their legal representative must understand the study and have voluntarily signed and dated the Informed Consent Form, which has been approved by the Sponsor and the Ethics Committee for this study.
3. Diagnosed with condition requiring surgical intervention per user manual.

   GLOW400 Specific Inclusion Criteria
4. Participants must have a suspected high-grade glioma (WHO grade III-IV) as evidenced by preoperative imaging modalities, which requires surgical intervention.
5. The active substance 5-aminolevulinic acid (5-ALA) fluorescence dye is administered according to the 5-ALA instructions for use.

   GLOW800 Specific Inclusion Criteria
6. Participants must have a condition requiring surgical intervention in the cerebral vascular area as well as during plastic and reconstructive surgery.
7. The Indocyanine Green (ICG) cyanine dye is administered as a contrast agent per instructions for use.

Candidates who meet any of the following exclusion criteria will not be eligible for recruitment in the study.

Exclusion Criteria:

1. Any uncontrolled systemic condition that may adversely affect the surgical outcome.
2. Individuals holding United States citizenship.

   GLOW400 Specific Exclusion Criteria
3. Known allergy to 5-ALA hydrochloride or protoporphyrin's.
4. Patients with porphyria (a condition characterized by the inability to break down protoporphyrin).

   GLOW800 Specific Exclusion Criteria
5. Known allergy to Indocyanine Green (ICG) cyanine dye.
6. Severe iodine-induced reactions to macromolecular iodine-containing compounds (e.g., iodinated contrast media, iodine-based antiseptics, or drugs like amiodarone), especially if the reaction involved anaphylaxis or respiratory compromise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended target population are patients undergoing a surgical procedure as defined within the intended purpose/indication for use of the respective compatible imaging system.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
White Light and Fluorescence image quality | Periprocedural
  Image quality will be assessed during surgery using a structured questionnaire completed by the operating surgeon. The evaluation includes white light and fluorescence imaging (GLOW400 and GLOW800) in both main surgeon (3D) and assistant (2D) modes. The following parameters will be rated:
  Contrast Color fidelity Stereoscopic/3D impression (main surgeon mode only) Resolution Latency (main surgeon mode only)
  Measurement Tool:
  MyVeo PMCF Study Data Collection Form - Questionnaire A and B
  Scale Range:
  5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent
  Interpretation of Scores:
  Scores of 3 or higher are considered acceptable. Ratings below 3 indicate performance concerns. The outcome will be analyzed using binary coding (Pass = 3-5; Fail = 1-2).

SECONDARY OUTCOMES:
The secondary objective will be assessed by evaluating the continued safety of the device by monitoring and analyzing adverse events, device-related complications. | Postprocedural
  Safety and User Experience will be evaluated using Questionnaire, completed postoperatively by the surgical team.
  It captures:
  Dizziness due to 3D visualization Surgical delays or interruptions Injuries to patient or user Breach of sterility Tissue burns
  Responses are binary for Safety:
  1. = Yes (event occurred)
  2. = No (event did not occur) Lower scores (2 = No) indicate better safety outcomes. The outcome is acceptable if no safety events are reported.
  User Experience
  It captures:
  1. ergonomics and comfort
  2. adjustability
  3. workflow
  4. confidence in terms of decision -making
  Each item is rated on a 5-point Likert scale:
  1. = Not available
  2. = Insufficient
  3. = Sufficient
  4. = Very good
  5. = Excellent Higher scores indicate better performance. The outcome is considered acceptable if all ratings are ≥3 (Sufficient or bett

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital Germans Trias I Pujol, Barcelona, Spain
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol